CLINICAL TRIAL: NCT03755453
Title: Assessment of Novel Measurement and Fitting Methods to Determine Their Reliability, Validity and Application
Brief Title: Assessment of Novel Measurement and Fitting Methods to Determine Their Reliability, Validity and Application - Sonova2018_34
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2018_34
Record Dates: First submitted 2018-09-28; First posted 2018-11-28 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: All participants will receive a hearing aid fitted with fitting method A and afterwards fitted with fitting method B.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audéo B-Direct fitted with fitting method A (Active Comparator): Traditional standard fitting method which do not include adjustments from the participants.
  Interventions: Device: Hearing aid: Phonak Audéo B90-Direct
- Audéo B-Direct fitted with fitting method B (Experimental): Alternative fitting method which includes additional adjustments from the participants.
  Interventions: Device: Hearing aid: Phonak Audéo B90-Direct

INTERVENTIONS:
Device: Hearing aid: Phonak Audéo B90-Direct — Hearing aids will be fitted to the participants individual hearing loss.

SUMMARY:
A methodical evaluation of novel measurement and fitting methods for individualizing CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired participants. The aim of the study is to investigate and asses strength and weaknesses of these novel measurement and fitting methods in terms of optimizing hearing performance and experience and/or usability of the hearing aids and accessories. Both laboratory measurements as well as evaluations in real life environments will be carried out. This will be a controlled and randomised active comparator clinical evaluation which will be conducted mono-centric at Sonova AG Headquarter based in Stäfa.

ELIGIBILITY:
Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Adult hearing impaired persons (minimum age: 18 years) with and without (experience with) hearing aids
* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Informed Consent as documented by signature

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend appointments
* Limited ability to describe listening impressions or to use hearing aids/ accessories
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of fitting method A versus B in regard to sound quality | 2 months
  The number of subjects who prefer the hearing aid setting achieved with hearing aid fitting method A versus B will be measured in the lab with the aid of sounds presented via loudspeakers. This will be measured with the Multiple Stimuli with Hidden Reference and Anchor (MUSHRA) method.

SECONDARY OUTCOMES:
Comparison of fitting method A versus B in regard to speech intelligibility in noise | 2 months
  The speech intelligibility in noise with hearing aid fitting method A versus B will be measured with the aid of the Oldenburg sentence test in dB Speech Reception Treshold (SRT).

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No